CLINICAL TRIAL: NCT02086682
Title: A Prospective Study of Airless Tubing in an Inpatient Acute Hemodialysis Unit in Hospitalized Patients in a Large Medical Center
Brief Title: A Prospective Study of Airless Tubing in an Inpatient Acute Hemodialysis Unit in Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: Marie Hogan (Other)
Collaborators: NxStage Medical (Other)
Responsible Party: Sponsor-Investigator, Marie Hogan, Associate Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Other Study IDs: 13-003161
Record Dates: First submitted 2014-03-10; First posted 2014-03-13 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-05

CONDITIONS: End Stage Renal Failure on Dialysis; Complication of Dialysis; Blood Coagulation Disorders
Keywords: hemodialysis; dialysis; renal dialysis; clotting; coagulation; blood lines
MeSH Terms: conditions — Blood Coagulation Disorders; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- General Care Cohort: The group included adult hospitalized patients requiring hemodialysis at the inpatient dialysis unit. This was an observational study, with no interventions.
- Critical Care Cohort: The group included adult hospitalized patients requiring hemodialysis at the intensive care unit. This was an observational study, with no interventions.

SUMMARY:
The introduction of unfractionated heparin (UFH), which prevents clotting of the extracorporal circuit, was one of the key advances that led to the rapid development and expansion of hemodialysis services. However, anticoagulation during hemodialysis of the patient at high risk for bleeding remains a frequently encountered problem in both inpatient and outpatient dialysis practice.

Streamline bloodlines are designed to eliminate blood-air contact. This is thought to help reduce heparin use and decrease clotting rates. The goal of this study was to prospectively examine impact of the Streamline airless blood tubing set, in an inpatient setting, on dialysis circuit clotting rates, anticoagulation use, and dialysis efficiency.

DETAILED DESCRIPTION:
The introduction of unfractionated heparin (UFH), which prevents clotting of the extracorporeal circuit, was one of the key advances that led to the rapid development and expansion of hemodialysis use, and remains the mainstay in hemodialysis practice today.

However, anticoagulation during hemodialysis of the patient at high risk for bleeding remains a frequently encountered problem in the nephrology practice. The need for anticoagulation to prevent clotting of the extracorporeal blood circuit and the need to prevent anticoagulation related bleeding complications in the patient has led to the development of numerous strategies; the safest from a bleeding standpoint being anticoagulant-free hemodialysis.

Streamline® bloodlines (Medisystems® Corporation, Lawrence, MA) are designed to eliminate blood-air contact. A pressure pod measures arterial and venous pressures without any blood-air contact. The venous chamber is run without an air gap. It is also designed so that blood flows in a circular vortex manner. This airless system is thought to provide several benefits: improved dialysis efficiency and blood flow rates, reduced heparin use and clotting rates.

The goal of this study was to prospectively examine the Streamline® airless tubing system in an inpatient setting and its association with clotting rates, and dialysis efficiency.

ELIGIBILITY:
Inclusion Criteria:

* All adult non-pregnant patients requiring inpatient hemodialysis at our center during the recruitment period until the target sample of dialysis sessions (n=1200) was reached.

Exclusion Criteria:

* Pregnant females
* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The group included adult hospitalized patients requiring hemodialysis at the inpatient dialysis unit or the ICU during the recruitment period.
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie C. Hogan, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Hospital, Saint Marys Campus, Rochester, Minnesota, United States

REFERENCES:
- [Result] Safadi S, Albright RC Jr, Dillon JJ, Williams AW, Alahdab F, Brown JK, Severson AL, Kremers WK, Ryan MA, Hogan MC. Prospective Study of Routine Heparin Avoidance Hemodialysis in a Tertiary Acute Care Inpatient Practice. Kidney Int Rep. 2017 Mar 16;2(4):695-704. doi: 10.1016/j.ekir.2017.03.003. eCollection 2017 Jul. PMID 29142987
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 338 patients were enrolled at the Mayo Clinic in Rochester, Minnesota from January 2014 to May 2015.
Period: Overall Study
Arm/Group | General Care Cohort | Critical Care Cohort
Started | 156 | 182
Completed | 156 | 182
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Care Cohort | Critical Care Cohort | Total
Number analyzed (Participants) | 156 | 182 | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (16) | 62 (17) | 62.5 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 67 | 127
  Male | 96 | 115 | 211
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 133 | 163 | 296
  More than one race | 0 | 7 | 7
  Unknown or Not Reported | 9 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United States | 156 | 182 | 338

OUTCOME MEASURES:

1. Primary Outcome: Clotting of Extracorporeal Dialysis Circuit
Description: Each dialysis session was prospectively observed for Clotting of Extracorporeal Dialysis Circuit. Events were defined as interruption of hemodialysis session, loss of the hemodialysis circuit, or inability to return blood to the patient upon rinse back.
Time Frame: During the dialysis session, approximately 211 minutes
Population: Units in the study referred to a dialysis session. A patient could have received dialysis more than once. Hence the number of patients (338) is less than the number of dialysis sessions (1200).
Measure: Number; unit: Clotting events
Units Other Than Participants: Dialysis Sessions
Arm/Group | General Care Cohort | Critical Care Cohort
Number analyzed (Participants) | 156 | 182
Number analyzed (Dialysis Sessions) | 600 | 600
Clotting events | 30 | 33
Statistical Analysis 1: Comparison: General Care Cohort vs Critical Care Cohort; Test type: Superiority; p = 0.79, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 30 days after hospital admission
Arm/Group | General Care Cohort | Critical Care Cohort
All-Cause Mortality (participants affected / at risk) | 31/156 | 40/182
Serious Adverse Events (participants affected / at risk) | 0/156 | 0/182
Other Adverse Events (participants affected / at risk) | 0/156 | 0/182

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No